CLINICAL TRIAL: NCT02747199
Title: Comparison Between SYNERGY™ vs. Bioresorbable Vascular Scaffold (BVS) ABSORB Neointimal Formation Assessed by (Optical Coherence Tomography) OCT and Coronary Angioscopy (CAS) Evaluation (The ENHANCE Study - ENdothelial Healing Assessment With Novel Coronary tEchnology)
Brief Title: ENdothelial Healing Assessment With Novel Coronary tEchnology
Acronym: ENHANCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Collaborators: Boston Scientific Corporation (Industry); Kurume University (Other)
Responsible Party: Principal Investigator, Wan Azman Wan Ahmad, Professor Dr, University of Malaya
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISROTH10249
Record Dates: First submitted 2016-04-19; First posted 2016-04-21 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Coronary Artery Disease
Keywords: SYNERGY; Neointimal formation; OCT; coronary angioscopy; coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Coronary artery implanted with SYNERGY stent (Active Comparator): One of the blocked coronary artery of a patient will received SYNERGY stent
  Interventions: Device: SYNERGY stent
- Coronary artery implanted with ABSORB scaffold (Active Comparator): Another blocked coronary artery of the same patient will received ABSORB scaffold
  Interventions: Device: BVS ABSORB scaffold

INTERVENTIONS:
Device: SYNERGY stent
  Arms: Coronary artery implanted with SYNERGY stent
Device: BVS ABSORB scaffold
  Arms: Coronary artery implanted with ABSORB scaffold

SUMMARY:
This is a prospective, non-randomized, single center clinical trial to assess neointimal coverage on the stent or scaffold strut and apposition of SYNERGY™ and ABSORB in minimum of 12 eligible human subject at 4 month and 12 month after stent or scaffold implantation using OCT and CAS

DETAILED DESCRIPTION:
All of the subject will received SYNERGY™ stent in one of the blocked coronary artery and ABSORB scaffold strut in the other artery. All subjects must have 2 coronary arteries stenosis of more than 70%.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 20 years old or older
2. Subject or legally authorized representative must provide written informed consent prior to any study related procedure, per site requirements.
3. Subject must have evidence of myocardial ischemia (eg stable or unstable angina, silent ischemia) suitable for elective PCI
4. Significant narrowing of at least 70% stenosis of de novo lesion (QCA or visual estimation) in 2 different native coronary arteries.
5. Subject is eligible for to undergo OCT and CAS examination at 4 months and 12 months after stent or scaffold implantation.
6. Subject is able to take dual anti-platelet therapy up to one year following the index procedure and anticoagulants prior/during the index procedure

Exclusion Criteria:

1. Subject had an acute myocardial infarction (STEMI or NSTEMI) within 24 hours of the index procedure
2. Subject has known left ventricular ejection fraction (LVEF) < 30%
3. Subject is receiving hemodialysis
4. Target vessel were treated by PCI within 12 months
5. Target lesion is located within a saphenous vein graft or an arterial graft
6. Target lesion is located in ostium
7. Target lesion is located highly tortuous equal to or greater than 60 degrees
8. Target lesion with TIMI flow 0 (total occlusion)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-08; Primary Completion 2016-07 (Actual); Study Completion 2017-04-12 (Actual)

PRIMARY OUTCOMES:
Apposition and neointimal coverage on the stent and scaffold strut | 4 months
  Neointimal coverage on the stent and scaffold strut and their apposition using OCT and CAS at 4 month after the stent implantation.

SECONDARY OUTCOMES:
Apposition and neointimal coverage on the stent and scaffold strut | 12 months
  Neointimal coverage on the stent or scaffold and their apposition using OCT and CAS at 12 month after stent implantation

CONTACTS AND LOCATIONS:
Overall Officials: Wan Azman Wan Ahmad, Principal Investigator — University Malaya Medical Center